CLINICAL TRIAL: NCT07342088
Title: The Combination of Lactobacillus Acidophilus DSMZ 26280 and Limosilolactobacillus Reuteri DSMZ 25441 Has an Impact on Clinical Course and Gut Microbiota of Children With Acute Infec-tious Diarrhea
Brief Title: Lactobacillus Acidophilus and Limosilactobacillus Reuteri for Acute Diarrhea in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Prof.Dr, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17042023126
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Infectious Diarrhea; Acute Gastroenteritis
Keywords: probiotic; acute infectious diarrhea; children; microbiota
MeSH Terms: conditions — Dysentery | interventions — Probiotics; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Probiotic combination of Lactobacillus acidophilus DSMZ 26280 (1×10⁸ CFU) and Limosilactobacillus reuteri DSMZ 25441 (1×10⁸ CFU), administered orally as drops once daily for 5 days, in addition to standard rehydration therapy.
  Interventions: Dietary Supplement: Probiotic; Other: Standard therapy
- Control group (Active Comparator): Standard therapy consisting of oral rehydration solution with or without intravenous fluids.
  Interventions: Other: Standard therapy

INTERVENTIONS:
Dietary Supplement: Probiotic — A probiotic preparation containing Lactobacillus acidophilus DSMZ 26280 (1×10⁸ CFU) and Limosilactobacillus reuteri DSMZ 25441 (1×10⁸ CFU) administered orally as drops once daily for 5 consecutive days, in addition to standard rehydration therapy.
  Arms: Probiotic Group
Other: Standard therapy — Standard management of acute infectious diarrhea consisting of oral rehydration solution with or without intravenous fluids according to clinical need.

SUMMARY:
This randomized controlled trial evaluated the effect of a combination of Lactobacillus acidophilus DSMZ 26280 and Limosilactobacillus reuteri DSMZ 25441 on the duration of diarrhea and gut microbiota composition in children aged 1-6 years with acute infectious diarrhea.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, open-label clinical trial was conducted between March 2024 and August 2024 at the Pediatric Emergency Department of Prof. Dr. İlhan Varank Sancaktepe Training and Research Hospital, Istanbul, Türkiye. Children aged 1-6 years presenting within 24 hours of onset of acute infectious diarrhea were randomized 1:1 to receive standard therapy (oral rehydration solution with or without intravenous fluids) alone or in combination with a probiotic preparation containing Lactobacillus acidophilus DSMZ 26280 (1×10⁸ CFU) and Limosilactobacillus reuteri DSMZ 25441 (1×10⁸ CFU) administered once daily for 5 days.

The primary outcomes were duration of diarrhea and the proportion of children who were diarrhea-free at 72 hours. Secondary outcomes included the proportion of children with diarrhea during the first 10 days of follow-up. A subgroup underwent longitudinal gut microbiota analysis at baseline, day 10, and day 30 using 16S rRNA sequencing.

The study was approved by the Ethics Committee of Prof. Dr. İlhan Varank Sancaktepe Training and Research Hospital (approval date April 17, 2024; decision no: 126), and written informed consent was obtained from all parents or legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-6 years
* Clinical diagnosis of acute infectious diarrhea
* Presentation within 24 hours of symptom onset
* Mild or no dehydration
* Written informed consent from parents or guardians

Exclusion Criteria:

* Antibiotic or probiotic use within the previous month
* Moderate or severe dehydration
* Malnutrition
* Immunosuppression
* Chronic systemic disease

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | Up to 10 days
  Time from randomization to last diarrheal stool
Proportion of children free of diarrhea at 72 hours | 72 hours after start of treatment
  Proportion of children free of diarrhea at 72 hours

SECONDARY OUTCOMES:
Proportion of children with ongoing diarrhea | Days 1-10
  Percentage of children with diarrhea recorded daily for the first 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Ilhan Varank Research and Training Hospital, University of Health Sciences,, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No